CLINICAL TRIAL: NCT03931720
Title: Clinical Research of ROBO1 Specific BiCAR-NK/T Cells on Patients With Malignant Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asclepius Technology Company Group (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AsclepiusTCG
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-tumor response of BiCAR-NK/T cells (ROBO1 CAR-NK/T cells) (Experimental): Patients with relapsed and refractory cancer of ROBO1 expression will be treated with BiCAR-NK/T cells (ROBO1 CAR-NK/T cells).
  Interventions: Biological: BiCAR-NK/T cells (ROBO1 CAR-NK/T cells)

INTERVENTIONS:
Biological: BiCAR-NK/T cells (ROBO1 CAR-NK/T cells) — The subject will be observed for any side effects during this time and all the adverse events will be recorded.

SUMMARY:
Immunotherapy has become the major breakthrough and the most promising treatment, with the host of development of tumor biology, molecular biology and immunology. ROBO1 is a potential target and spectacular paradigm in the diagnosis and treatment of solid tumors. This study is for evaluation of the safety and efficacy of ROBO1 CAR-NK/T cell immunotherapy for malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~75 years old, male or female
2. Life expectancy ≥ 6 months
3. ECOG score: 0-3
4. ROBO1 expression in malignancy tissues detected by immuno-histochemistry (IHC)
5. Advanced solid tumor was diagnosed by pathological or clinical physicians
6. Laboratory examination: white blood cell≥3 x 10*9/L, blood platelet count≥70 x 10*9/L, hemoglobin≥80g/L, lymphocyte count≥15%, total bilirubin≤100 mol/L, ALT and AST less than five times of the normal level, serum creatinine less than 1.5 times of the normal level
7. Signed informed consent
8. Women of child-bearing age must have evidence of negative pregnancy test and be willing to practice birth control after 2 weeks following the cell transfusion

Exclusion Criteria:

1. Expected overall survival < 6 months
2. Patients with uncontrolled hypertension, unstable coronary disease (uncontrolled arrhythmias, unstable angina, decompensated congestive heart failure (> Class II, NYHA), or myocardial infarction within 6 months
3. Abnormal lung function: FEV (forced expiratory volume) < 30% prediction, DLCO (diffusing capacity of the lung for carbon monoxide) < 30% prediction, blood oxygen saturation < 90%
4. Other serious diseases: nervous, mental disorders, immune regulatory diseases, metabolic diseases, infectious diseases, etc.
5. Unable or unwilling to provide informed consent, or fail to comply with the test requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events as assessed by CTCAE v4.03 | 1 year
  Defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Suzhou Kowloon Hospital, Shanghai Jiaotong University School of Medicine, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No